CLINICAL TRIAL: NCT00245076
Title: Evaluation of the Impact of a Bulletin Board on a Web-Based Smoking Cessation Intervention
Brief Title: Smokefree.Gov Website in Helping United States Federal Employees Quit Smoking
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Masking: None | Purpose: Prevention
Other Study IDs: CDR0000450773; TCRB-OHSR-2765
Record Dates: First submitted 2005-10-25; First posted 2005-10-27 (Estimated); Last update posted 2015-05-01 (Estimated); Status verified 2006-04

CONDITIONS: Unspecified Adult Solid Tumor, Protocol Specific
Keywords: unspecified adult solid tumor, protocol specific

INTERVENTIONS:
Behavioral: smoking cessation intervention
Other: internet-based intervention

SUMMARY:
RATIONALE: Stop-smoking information on the smokefree.gov website may help people quit smoking and remain a nonsmoker.

PURPOSE: This clinical trial is studying how well the smokefree.gov website works with an electronic bulletin board in helping United States federal employees quit smoking.

DETAILED DESCRIPTION:
OBJECTIVES:

* Determine the perception of utility of the current, publicly accessible version of the smokefree.gov website and the addition of an electronic bulletin board and its features, including open-ended comments, in promoting smoking cessation among United States federal employees who are currently smokers.
* Determine the use of this tool, in terms of average length of time spent on the website, number of page clicks, most popular page clicks, and key interest areas, among these participants.
* Determine the changes in smoking habits, in terms of smoking reduction and short- and long-term abstinence, among these participants.

OUTLINE: This is an open-label study.

Participants are encouraged to use the smokefree.gov website as frequently as needed for support and resources while trying to quit smoking and become, and remain, nonsmokers. Participants are invited to provide feedback on the usefulness of self-help guidelines and several other tools. Participants complete questionnaires evaluating the website at study entry and at 1, 3, and 6 months after study entry.

PROJECTED ACCRUAL: A total of 4,200 participants will be accrued for this study.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Currently smokes > 1 cigarette daily by self reporting
* Planning to quit smoking in the next 90 days by self reporting
* Must be a federal employee or federally employed

PATIENT CHARACTERISTICS:

Performance status

* Not specified

Life expectancy

* Not specified

Hematopoietic

* Not specified

Hepatic

* Not specified

Renal

* Not specified

PRIOR CONCURRENT THERAPY: Any prior or concurrent therapy allowed

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Dates: Start 2005-04; Study Completion 2007-10 (Actual)

PRIMARY OUTCOMES:
Abstinence for 7 consecutive days and 24 hours at 1, 3, and 6 months

SECONDARY OUTCOMES:
Visits to the website after registration at 1, 3, and 6 months
Satisfaction with the website at 1, 3, and 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Jacqueline Stoddard, PhD, MA, Principal Investigator — National Cancer Institute (NCI)
Locations (1):
- Tobacco Control Research Branch, Rockville, Maryland, United States

REFERENCES:
- [Derived] Stoddard JL, Augustson EM, Moser RP. Effect of adding a virtual community (bulletin board) to smokefree.gov: randomized controlled trial. J Med Internet Res. 2008 Dec 19;10(5):e53. doi: 10.2196/jmir.1124. PMID 19097974